CLINICAL TRIAL: NCT05104320
Title: A Partially Randomized Patient Preference Trial to Assess the Quality of Life and Patency Rate After Minimally Invasive Cardiac Surgery-Coronary Artery Bypass Grafting: the MICS-CABG PRPP Trial
Brief Title: The Quality of Life and Patency Rate After Minimally Invasive Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU MICS-CABG PRPP Trial
Record Dates: First submitted 2021-10-09; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-09

CONDITIONS: Minimally Invasive Cardiac Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MICS-CABG (Experimental): Patients undergoing MICS-CABG.
  Interventions: Procedure: MICS-CABG
- sternotomy CABG (Active Comparator): Patients undergoing thoracotomy OPCABG.
  Interventions: Procedure: sternotomy CABG

INTERVENTIONS:
Procedure: MICS-CABG — Off-pump multi-vessel coronary artery bypass grafting via left thoracotomy under minimally invasive conditions.
  Arms: MICS-CABG
Procedure: sternotomy CABG — Off-pump multi-vessel coronary artery bypass grafting with conventional thoracotomy.
  Arms: sternotomy CABG

SUMMARY:
This trial will address essential questions of the efficacy and safety of MICS-CABG in addition to the quality of life and patency rate of the grafts. The study will also address the impact of patients' preferences on external validity and internal validity.

In this study, patients with a preference will be allocated to treatment strategies accordingly, whereas only those patients without a distinct preference will be randomized. The randomized trial is a 248-patient controlled, randomized, investigator-blinded trial. It is designed to compare whether treatment with MICS-CABG is beneficial in comparison to CABG. This study is aimed to establish the superiority hypothesis for the physical component summary (PCS) accompanied by the noninferiority hypothesis for overall graft patency. Patients with no treatment preference will be randomized in a 1:1 fashion to one of the two treatment arms.

The primary efficacy endpoints are the PCS score at 30 days after surgery and the overall patency rate of the grafts within 14 days after surgery. Secondary outcome measures include the PCS score and patency rate at different time points. Safety endpoints include major adverse cardiac and cerebrovascular events, complications, bleeding, wound infection, death, etc.

ELIGIBILITY:
Inclusion Criteria:(A patient will be included in the study when the following criteria and requirements are met)

① Patient age of ≥25 years but ≤85 years, and patients with CAD who require multivessel coronary bypass surgery. ② Angina that affects daily life and work and is uncontrollable with conservative treatment. ③ Significant stenosis in the left main (LM) coronary artery, left anterior descending (LAD) branch or left circumflex (LCX) branch >70%. ④ Severe stenosis (stenosis degree >75%) of three main branches of the coronary artery (anterior descending branch, circumflex branch, right coronary artery) with the need to undergo off-pump coronary artery bypass surgery.

Exclusion Criteria:(A patient will be excluded from the study if they meet any of the following criteria)

① Unstable preoperative hemodynamic status (vasoactive drugs such as dopamine, epinephrine or norepinephrine to maintain blood pressure, or an intra-aortic balloon pump [IABP] is implanted preoperatively) or requiring emergency surgery. ② Severe emphysema, hypoxemia [postbronchodilator forced expiratory volume in 1 s (FEV1)/forced vital capacity (FVC)<70% and FEV1% predicted<50% or partial pressure of oxygen (pO2)<60 mmHg or partial pressure of carbon dioxide (pCO2)>40 mmHg without oxygen therapy. ③ Old extensive myocardial infarction without a viable myocardium based on isotope and echocardiography examination, significant cardiac enlargement (cardiothoracic ratio>0.75, EF<30%, left ventricular diastolic diameter (LVDd)>60 mm, left ventricular aneurysm or severe arrhythmia). ④ Severe pleural adhesion, chest deformity, or previous thoracic radiotherapy. ⑤Previous thoracotomy surgery. ⑥ Simultaneous valve or other cardiac surgery. ⑦Planned cardiopulmonary bypass surgery. ⑧Poor condition of the distal coronary artery (diffuse stenosis, chronic total obstructive lesion with severe calcification or inability to match the graft due to a small diameter (<1.0 mm). ⑨Intolerance to surgery in combination with the following complications: Terminal cancer, uncontrolled infection, bleeding, severe brain injury, infarction or bleeding, multiple organ failure and other major organ dysfunction such as severe liver dysfunction or severe congestive heart failure.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2021-10-31 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
SF-36 PCS score | 30 days after surgery
  The SF-36 is a concise health test that features Physical Functioning (PF), Roe-Physical (RP), Bodily Pain, General Health (GH), Vitality (VT), Social Functioning (SF), Roe-Emotional (Emotional) and Mental Health (MH) functioning and comprehensively summarizes the quality of life of the respondents across 8 aspects. The PCS and mental component summary (MCS) can be calculated from the eight abovementioned indicators with different weights. The PCS and the MCS each range from 0 to 50, with a lower score indicating worse quality of life (QoL) and a higher score indicating better QoL.
Overall patency rate of the grafts | within 14 days after surgery
  the patency rates of the LIMA, RIMA, saphenous vein graft (SVG) and radial artery (RA) will be evaluated by the Fitzgibbon A+B grade

SECONDARY OUTCOMES:
SF-36 PCS scores | 7 days, 3 months, 6 months and 1 year after surgery
  The SF-36 is a concise health test that features Physical Functioning (PF), Roe-Physical (RP), Bodily Pain, General Health (GH), Vitality (VT), Social Functioning (SF), Roe-Emotional (Emotional) and Mental Health (MH) functioning and comprehensively summarizes the quality of life of the respondents across 8 aspects. The PCS and mental component summary (MCS) can be calculated from the eight abovementioned indicators with different weights. The PCS and the MCS each range from 0 to 50, with a lower score indicating worse quality of life (QoL) and a higher score indicating better QoL.
SF-36 MCS scores | 7 days, 3 months, 6 months and 1 year after surgery
  The SF-36 is a concise health test that features Physical Functioning (PF), Roe-Physical (RP), Bodily Pain, General Health (GH), Vitality (VT), Social Functioning (SF), Roe-Emotional (Emotional) and Mental Health (MH) functioning and comprehensively summarizes the quality of life of the respondents across 8 aspects. The PCS and mental component summary (MCS) can be calculated from the eight abovementioned indicators with different weights. The PCS and the MCS each range from 0 to 50, with a lower score indicating worse quality of life (QoL) and a higher score indicating better QoL.
Patency rate of the different material grafts | 14 days and 1 year after surgery
  the patency rates of the LIMA, RIMA, saphenous vein graft (SVG) and radial artery (RA) will be evaluated by the Fitzgibbon A+B grade
Length of incubation | within 7 days after surgery
  the time of assisted respiratory ventilation after surgery
Hospitalization cost | within 7 days after surgery
  total hospitalization cost of each patient
Length of postoperative hospitalization time | within 7 days after surgery
  total postoperative hospitalization time of the patients
Bypass surgical variation index | within 7 days after surgery
  The actual graft number is compared with the preoperative strategy. If the actual number of grafts is less than that in the preoperative plan, the results will be recorded.
Intrahospital RBC transfusion volume | within 7 days after surgery
  the amount of red blood cells (U) to be transfused during hospitalization. Indications for blood transfusion include hemoglobin less than 90 g/L, severe intraoperative or postoperative active bleeding, or other blood transfusion considered necessary by the surgeons.
Wound infection rate | within 3 months after surgery
  wound dehiscence, effusion and secondary debridement and suture
Number of Participants with re-exploration for bleeding or other causes (not including wound-related causes) | within 1 year after surgery
  the requirement to return to the operating room for reopening of sternotomy or MICS CABG incision for any reason, such as bleeding, postoperative acute myocardial ischemia and unexplained circulatory instability. Debridement for DSWI or infection of anterior-lateral wounds will be excluded.
Major adverse cardiac and cerebrovascular events (MACCEs) | 1, 6, 12, 24, 36, and 60 months after surgery
  Composite endpoint of all-cause death, nonfatal myocardial infarction, stroke, and target vessel ischemia-driven repeated revascularization (TVR).

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Ling, Study Chair — Peking University Third Hospital; Yichen Gong, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT05104320/Prot_SAP_000.pdf